CLINICAL TRIAL: NCT05025111
Title: Entia Liberty: Clinical Performance Validation - Capillary Performance
Brief Title: Entia Liberty: Capillary Validation
Status: Completed | Type: Observational
Sponsor: Entia Ltd (Industry)
Collaborators: The Christie NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 304718
Record Dates: First submitted 2021-08-26; First posted 2021-08-27 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Entia Liberty — Home monitoring device

SUMMARY:
This study is a clinical performance validation study to evaluate the performance of the Entia Liberty device. Patients undergoing routine venepuncture blood tests will be recruited to have an Entia Liberty test (by finger-prick) done on them by a trained healthcare professional. The results from that finger-prick test will be compared against the results from the routine venepuncture blood test (reference method) and subsequently, excess blood from the routine venepuncture test will be run on another Entia Liberty device in the laboratory. All three results (Entia Liberty capillary, Entia Liberty venous and gold standard venous) will be compared against each other to prove Entia Liberty's performance claims.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old at the time of study entry
* Currently receiving standard of care systemic anti- cancer therapy (chemotherapy, immunotherapy, endocrine and targeted therapy) for solid organ malignancy and has received at least one cycle.
* Scheduled to be undergoing routine venous laboratory blood tests as part of standard of care
* Can provide written informed consent
* Blood samples collected and stored in K2-EDTA vacutainers only

Exclusion Criteria:

* Known inherited or acquired bleeding disorder
* History of haematological malignancy
* Known poorly controlled anti-coagulation
* Inadequate use and understanding of the English language, requiring a translator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be recruited from the outpatients clinic at the Christie, while they are waiting for their blood tests.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-09-12 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
To obtain/validate the value of the total error of the Entia Liberty device. | 3 months
  The dataset from this study will provide evidence to support the device's performance claims.
To obtain/validate the value of the linearity of the Entia Liberty device. | 3 months
  The dataset from this study will provide evidence to support the device's performance claims.
To obtain/validate the value of the bias of the Entia Liberty device. | 3 months
  The dataset from this study will provide evidence to support the device's performance claims.

CONTACTS AND LOCATIONS:
Locations (2):
- United Kingdom (2):
  - The Christie NHS Foundation Trust, Manchester
  - Royal Albert Edward Infirmary, Wigan